CLINICAL TRIAL: NCT04474197
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled Study of the Efficacy and Safety of VX-864 in PiZZ Subjects
Brief Title: Evaluation of the Efficacy and Safety of VX-864 in Subjects With the PiZZ Genotype
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX19-864-101; 2019-004881-16 (EudraCT Number)
Record Dates: First submitted 2020-07-13; First posted 2020-07-16 (Actual); Results first posted 2022-05-26 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Alpha1-Antitrypsin Deficiency
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Participants received placebo matched to VX-864 in the treatment period for 28 days.
  Interventions: Drug: Placebo
- VX-864 100 mg (Experimental): Participants received VX-864 100 milligrams (mg) every 12 hours (q12h) in the treatment period for 28 days.
  Interventions: Drug: VX-864
- VX-864 300 mg (Experimental): Participants received VX-864 300 mg q12h in the treatment period for 28 days.
  Interventions: Drug: VX-864
- VX-864 500 mg (Experimental): Participants received VX-864 500 mg q12h in the treatment period for 28 days.
  Interventions: Drug: VX-864

INTERVENTIONS:
Drug: VX-864 — Tablets for oral administration.
  Arms: VX-864 100 mg; VX-864 300 mg; VX-864 500 mg
Drug: Placebo — Placebo matched to VX-864 for oral administration.
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy, safety and pharmacokinetics (PK) of VX-864 in PiZZ subjects.

ELIGIBILITY:
Key Inclusion Criteria:

* Subjects must have a PiZZ genotype confirmed at screening
* Plasma AAT levels indicating severe deficiency at screening

Key Exclusion Criteria:

* History of a medical condition that could negatively impact the ability to complete the study
* Solid organ, or hematological transplantation or is currently on a transplant list
* History of use of gene therapy or RNAi therapy at any time previously

Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2020-07-24 (Actual); Primary Completion 2021-05-04 (Actual); Study Completion 2021-05-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (30):
- United States (22):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - University of California Davis Medical Center, Sacramento, California
  - National Jewish Health, Denver, Colorado
  - University of Florida, Gainesville, Florida
  - University of Miami Miller School of Medicine, Miami, Florida
  - Central Florida Pulmonary, Orlando, Florida
  - The University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Minnesota, Minneapolis, Minnesota
  - Blessing Corporate Services, Inc., dba Blessing Health System, Hannibal, Missouri
  - Cardinal Glennon Children's Hospital - St. Louis University, St Louis, Missouri
  - University of North Carolina Medical Center, Chapel Hill, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Renovatio Clinical, Houston, Texas
  - The University of Texas Health Science Center at Tyler, Tyler, Texas
  - University of Utah Health, Salt Lake City, Utah
  - Inova Fairfax Medical Campus, Falls Church, Virginia
- Canada (2):
  - Queen Elizabeth II Health Sciences Center, Halifax
  - Inspiration Research Ltd, Toronto
- Germany (3):
  - University Hospital RWTH Aachen, Aachen
  - Universitätsklinikum Essen, Essen
  - Medizinische Hochschule Hannover, Hanover
- Royal College of Surgeons in Ireland Clinical Research Centre, Beaumont Hospital, Beaumont, Ireland
- Skanes Universitetssjukhus, Malmo, Malmo, Sweden
- Staploe Medical Centre, Soham Ely, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was conducted in participants 18 through 80 of years of age, inclusive with the PiZZ genotype.
Period: Overall Study
Arm/Group | Placebo | VX-864 100 mg | VX-864 300 mg | VX-864 500 mg
Started | 7 | 10 | 9 | 18
Completed | 7 | 9 | 9 | 18
Not Completed | 0 | 1 | 0 | 0
Not completed — Withdrawal of consent (not due to adverse event) | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- VX-864 100 mg: Participants received VX-864 100 mg q12h in the treatment period for 28 days.
- Total: Total of all reporting groups
Arm/Group | Placebo | VX-864 100 mg | VX-864 300 mg | VX-864 500 mg | Total
Number analyzed (Participants) | 7 | 10 | 9 | 18 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (10.5) | 55.1 (5.3) | 53.2 (16.2) | 57.4 (9.9) | 57.0 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 6 | 14 | 31
  Male | 2 | 4 | 3 | 4 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 7 | 8 | 8 | 15 | 38
  Unknown or Not Reported | 0 | 2 | 1 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 7 | 10 | 9 | 18 | 44
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Plasma Functional Alpha-1 Antitrypsin (AAT) Levels [Mean (Standard Deviation); unit: micromole per liter] | 4.7 (1.3) | 4.0 (0.7) | 3.8 (0.9) | 4.1 (0.6) | 4.1 (0.9)

OUTCOME MEASURES:

1. Primary Outcome: Change in Plasma Functional Alpha-1 Antitrypsin (AAT) Levels
Time Frame: From Baseline at Day 28
Population: Full analysis set (FAS) included all randomized participants who received at least 1 dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: micromole per liter
Groups:
- VX-864 300 mg: Participants received VX-864 300 mg dose q12h in the treatment period for 28 days.
- VX-864 500 mg: Participants received VX-864 500 mg dose q12h in the treatment period for 28 days.
Arm/Group | Placebo | VX-864 100 mg | VX-864 300 mg | VX-864 500 mg
Number analyzed (Participants) | 7 | 10 | 9 | 18
micromole per liter | -0.1 (0.3) | 2.3 (0.3) | 2.3 (0.2) | 2.1 (0.2)
Statistical Analysis 1: Comparison: Placebo vs VX-864 100 mg; Test type: Superiority; p < 0.0001, Mixed-effects Model for Repeated Measure; Least Squares (LS) Mean Difference = 2.3, 95% CI 2-sided [1.5 to 3.1]
Statistical Analysis 2: Comparison: Placebo vs VX-864 300 mg; Test type: Superiority; p < 0.0001, Mixed-effects Model for Repeated Measure; LS Mean Difference = 2.3, 95% CI 2-sided [1.6 to 3.1]
Statistical Analysis 3: Comparison: Placebo vs VX-864 500 mg; Test type: Superiority; p < 0.0001, Mixed-effects Model for Repeated Measure; LS Mean Difference = 2.2, 95% CI 2-sided [1.5 to 2.9]

2. Primary Outcome: Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Time Frame: Day 1 up to Week 8
Population: The safety set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo | VX-864 100 mg | VX-864 300 mg | VX-864 500 mg
Number analyzed (Participants) | 7 | 10 | 9 | 18
participants
  Participants With AEs | 4 | 7 | 7 | 17
  Participants With SAEs | 0 | 0 | 0 | 2

3. Secondary Outcome: Change in Plasma Antigenic AAT Levels
Time Frame: From Baseline at Day 28
Population: FAS.
Measure: Least Squares Mean (Standard Error); unit: micromole per liter
Arm/Group | Placebo | VX-864 100 mg | VX-864 300 mg | VX-864 500 mg
Number analyzed (Participants) | 7 | 10 | 9 | 18
micromole per liter | -0.1 (0.4) | 3.4 (0.4) | 2.9 (0.4) | 2.6 (0.2)
Statistical Analysis 1: Comparison: Placebo vs VX-864 100 mg; Test type: Superiority; p < 0.0001, Mixed-effects Model for Repeated Measure; LS Mean Difference = 3.5, 95% CI 2-sided [2.4 to 4.6]
Statistical Analysis 2: Comparison: Placebo vs VX-864 300 mg; Test type: Superiority; p < 0.0001, Mixed-effects Model for Repeated Measure; LS Mean Difference = 3.0, 95% CI 2-sided [1.9 to 4.0]
Statistical Analysis 3: Comparison: Placebo vs VX-864 500 mg; Test type: Superiority; p < 0.0001, Mixed-effects Model for Repeated Measure; LS Mean Difference = 2.7, 95% CI 2-sided [1.8 to 3.7]

4. Secondary Outcome: Observed Pre-dose Plasma Concentration (Ctrough) of VX-864
Time Frame: Pre-dose at Day 7, Day 14, Day 21 and Day 28
Population: Pharmacokinetic (PK) set included participants who received at least 1 dose of study drug. Here "Number analyzed" signifies those participants who were evaluable for this endpoint at specified time points.
Measure: Mean (Standard Deviation); unit: microgram per milliliter
Arm/Group | VX-864 100 mg | VX-864 300 mg | VX-864 500 mg
Number analyzed (Participants) | 10 | 9 | 18
microgram per milliliter
  Day 7: number analyzed (Participants) | 9 | 8 | 16
  Day 7 | 1.13 (0.743) | 1.62 (0.665) | 2.74 (2.89)
  Day 14: number analyzed (Participants) | 8 | 9 | 18
  Day 14 | 0.852 (0.340) | 1.47 (0.847) | 4.35 (5.36)
  Day 21: number analyzed (Participants) | 8 | 8 | 18
  Day 21 | 0.868 (0.503) | 1.21 (0.770) | 1.79 (0.922)
  Day 28: number analyzed (Participants) | 9 | 8 | 18
  Day 28 | 0.797 (0.327) | 1.29 (0.646) | 2.55 (2.40)

ADVERSE EVENTS:
Time Frame: Day 1 up to Week 8
Arm/Group | Placebo | VX-864 100 mg | VX-864 300 mg | VX-864 500 mg
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/10 | 0/9 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/10 | 0/9 | 2/18
Other Adverse Events (participants affected / at risk) | 4/7 | 7/10 | 7/9 | 17/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=7) | VX-864 100 mg (N=10) | VX-864 300 mg (N=9) | VX-864 500 mg (N=18)
Chest pain (General disorders) | 0 | 0 | 0 | 1
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=7) | VX-864 100 mg (N=10) | VX-864 300 mg (N=9) | VX-864 500 mg (N=18)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Eye allergy (Eye disorders) | 0 | 0 | 0 | 1
Macular degeneration (Eye disorders) | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 4
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 2 | 4
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 2 | 0 | 3
Feeling abnormal (General disorders) | 0 | 1 | 0 | 0
Feeling cold (General disorders) | 0 | 1 | 0 | 1
Malaise (General disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 2 | 1 | 0
Infective exacerbation of bronchiectasis (Infections and infestations) | 0 | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 1
Back injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Post procedural contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Vaccination complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Blood bicarbonate decreased (Investigations) | 0 | 0 | 1 | 0
Blood cholesterol increased (Investigations) | 1 | 0 | 1 | 1
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 1
Blood pressure diastolic increased (Investigations) | 0 | 0 | 0 | 1
Blood triglycerides increased (Investigations) | 0 | 0 | 1 | 1
Haemoglobin increased (Investigations) | 0 | 1 | 0 | 1
Low density lipoprotein increased (Investigations) | 1 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 1 | 0
Oxygen saturation decreased (Investigations) | 0 | 1 | 0 | 0
Protein total decreased (Investigations) | 0 | 0 | 0 | 1
Red blood cell count increased (Investigations) | 0 | 0 | 0 | 1
White blood cells urine positive (Investigations) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 2 | 1
Dysaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 2 | 2
Tremor (Nervous system disorders) | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1
Poor quality sleep (Psychiatric disorders) | 0 | 0 | 0 | 1
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Polymorphic light eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-01-12): https://cdn.clinicaltrials.gov/large-docs/97/NCT04474197/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-11): https://cdn.clinicaltrials.gov/large-docs/97/NCT04474197/SAP_001.pdf